CLINICAL TRIAL: NCT03329924
Title: ICU Liberation: Does Enhanced Patient Mobilization Improve Outcomes?
Status: Completed | Type: Observational
Sponsor: Bassett Healthcare (Other)
Responsible Party: Principal Investigator, Erik Riesenfeld, Attending Physician - Critical Care & Pulmonology, Bassett Healthcare
Other Study IDs: 2084
Record Dates: First submitted 2017-10-31; First posted 2017-11-06 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Early Mobilization of Mechanically Ventilated Patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pre-implementation cohort: These patients are being exposed to the current standard of care, which does include some early mobilization practices, but not a formalized program.
  Interventions: Other: Activity level measurement by accelerometer
- post-implementation cohort: These patients will have been exposed to the fully executed early mobilization program.
  Interventions: Other: Activity level measurement by accelerometer

INTERVENTIONS:
Other: Activity level measurement by accelerometer — Eligible patients will wear an accelerometer to measure activity levels while in the ICU.

SUMMARY:
The hypothesis of this study is that an early mobilization program coupled with organizational efforts to implement the ABCDEF bundle will increase the rate of ICU patient mobilization and decrease the ICU length of stay, but will not significantly affect patient mortality. Mobilization efforts will be done to improve patient care and the study will allow for measurement of the effects of implementation of this effort. The early mobilization program is being instituted as standard of care. The study will measure the actual degree of change in patients' activity level and to evaluate the effect of the program on outcome measures such as length of stay.

DETAILED DESCRIPTION:
The purpose of this study is to study implementation efficacy of an early mobilization program in a rural mixed surgical and medical ICU.

The aim of the study is to test whether a program of early mobilization training along with ongoing ABCEDF bundle implementation will change the following:

1. early mobilization of ventilated patients in the ICU measured using accelerometer data as a primary measure along with other nurse reported data from the EMR
2. ICU length of stay
3. other clinical variable outlined in the design section

This study will have a pre- and post-implementation design. Baseline activity levels of eligible patients will be collected prospectively for approximately 3 months while staff is being trained and the details of the early mobilization program are being finalized. All eligible patients will wear an accelerometer while in the ICU. Length of ICU stay, total hospitalization, discharge disposition, and the occurrence of certain hospital-acquired complications will also be recorded as part of the baseline/current practice data. There will be a pause in data collection as the early mobilization program is incorporated into standard practice.

Data collection will resume approximately one month after the implementation of the program.

All eligible patients will wear an accelerometer to measure activity level while in the ICU. Length of ICU stay, total hospitalization, discharge disposition, and the occurrence of certain hospital-acquired complications will also be recorded. Other variables to be assessed include: ICU staffing costs, overall hospitalization costs, rate of patient falls, rate of staff injuries, level of exercise tolerance achieved by time of discharge.

ELIGIBILITY:
Inclusion Criteria:

* - Patients in a rural mixed surgical and medical ICU requiring mechanical ventilation

Exclusion Criteria:

* age less than 18
* Pregnant patients
* Cardiac surgery patients
* "boarding" patients in the ICU
* Patients expected to be extubated in less than 24 total hours (e.g. combative trauma patient intubated in order to complete workup),
* Patients unable to walk prior to admission
* Patients without limbs
* Patients with an unstable spinal injury.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in a rural mixed surgical and medical ICU requiring mechanical ventilation will be included in this study
Sampling Method: Non-Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Activity level | one week
  activity level during a patient's ICU admission will be measured by accelerometer

SECONDARY OUTCOMES:
Length of ICU admission | one week
  the amount of time spent as as an admitted patient to the ICU will be measured
length of total hospitalization | one month
  the total amount of time spent as an inpatient for this episode of care will be measured

CONTACTS AND LOCATIONS:
Overall Officials: Erik riesenfeld, MD, Principal Investigator — Bassett Medical Center
Locations (1):
- Bassett Medical Center, Cooperstown, New York, United States

IPD SHARING:
Plan to Share IPD: No